CLINICAL TRIAL: NCT03267927
Title: Management of Obstructive Sleep Apnea (OSA) in Children and Maxillary and Mandibular Development
Acronym: SAOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 35RC16_9851_SAOS
Record Dates: First submitted 2017-08-28; First posted 2017-08-31 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: OSA; Polysomnography; Rapid palatal expansion; Mandibular advancement; Sleep position
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with OSA (Experimental)
  Interventions: Device: Rapid palatal expansion; Device: MGA™ system; Device: Yoobreath™ system

INTERVENTIONS:
Device: Rapid palatal expansion — Fixation of rapid palatal expansion from day 0 to day 60
Device: MGA™ system — Use of a mandibular advancement Appliance during the night from day 60 to day 180 (end of treatment from day 120 if Angle Class I is obtained)
Device: Yoobreath™ system — Use of a device allowing sleep in a semi-seated position during the night from day 15 to day 180 (end of treatment from day 120 if Angle Class I is obtained)

SUMMARY:
Assessment of the association of maxillary expansion using a rapid palatal expansion, use of a mandibular advancement appliance (MGA™) and of a device allowing sleep in a semi-seated position (Yoobreath™) in patients with Obstructive Sleep Apnea (OAS). MGA™ and YooBreath™ constitute the Yookid system™.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea syndrome (OSA) shows a 10% morbidity rate in children with a higher rate between the ages of 3 and 5. Generally speaking, its prevalence is underestimated. Furthermore, detecting OSA remains difficult due to its particular physiopathology. The decrease in nasopharyngeal airway dimensions is the most common etiology. This decrease is related to soft tissues as well as maxillomandibular abnormalities. The aim of the study is to show that reducing sleep apnea in children remains possible when inducing rapid palatal expansion and mandibular advancement using the Yookid™ system. The Yookid™ system associates a mandibular advancement appliance and repositioning of the patient during sleep.

ELIGIBILITY:
Inclusion Criteria:

* 5 to 7 year-old children
* Children with American Society of Anesthesiologists score (ASA) of 1 and 2
* Children with signs of OSA during examination and clinical exam
* Children with apnea-hypopnea index (AHI) from 1 to 5 (one to five sleep apnea / hour during PSG)
* Children with a class II division 1 angle malocclusion (at the canines level rotation center) and skeletal class II according to Delaire analysis

Exclusion Criteria:

* OSA associated to syndromic disorder and/or syndrome
* Body/Mass Index (BMI) > 97ème percentile according to development curves (obese children)
* Central sleep apnea
* Respiratory allergy
* Previous ear, nose and throat (ENT) surgery
* Hypertrophic tonsils needing surgery
* Adenoid hypertrophy needing surgery
* Patients with ankyloglossia

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2017-11-05 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

PRIMARY OUTCOMES:
Assessment in 5 to 7 year-old children the efficacy on OSA (removal or decrease of apnea/hypopnea) of Rapid Palatal Expansion combined with advancement using a mandibular advancement appliance (MGA™) | Day 180
Assessment in 5 to 7 year-old children the efficacy on OSA (removal or decrease of apnea/hypopnea) of Rapid Palatal Expansion combined with a device allowing a semi-seated sleeping position (YooBreath™) | Day 180

SECONDARY OUTCOMES:
Sleep improvement | Day -7, day 180
  Measurement by polysomnography of desaturation index, micro arousal index and snoring index
Assessment of quality of sleep | Day 180
  Assessment of quality of sleep by a questionnaire
Assessment of quality of wakefulness | Day 180
  Assessment of quality of wakefulness by a questionnaire
Measurement of lengthening of mandibular body and ramus | Day -7, day 180
  Assessment of mandible development by an orthodontist using cephalometric analysis
Improvement of breathing | Day -7, day 180
  Improvement of breathing defined by polysomnography
Assessment of dental occlusion | Day -7, day 180
  Assessment of dental occlusion (clinical and using casts): diagnosis of Angle class
Assessement by the child and the parents of the treatment and the devices used | Day 180
  Assessement by the child and the parents of the treatment and the devices used by two questionnaires (one for parents and one for the child)
Assessment of intensity of pain during rapid palatal expansion | Day 60
  Assessment of intensity of pain after fixing of rapid palatal expansion using a Visual Analogue Scale (VAS)
Assessment of duration of pain during rapid palatal expansion | Day 60
  Number of painful days after fixing of rapid palatal expansion
Assessment of intensity of dental pain the morning on waking after using the MGA™ system | Day 60, day 90, day 120, day 150, day 180
  Assessment of intensity of dental pain the morning on waking using a Visual Analogue Scale (VAS)
Assessment of salivary disorders the morning on waking after using the MGA™ system | Day 60, day 90, day 120, day 150, day 180
  Assessment of salivary disorders the morning on waking by a questionnaire
Assessment of duration of dental pain the morning on waking after using the MGA™ system | Day 60, day 90, day 120, day 150, day 180
  Number of painful days at the mandible the morning on waking
Assessment of pain related to the semi-seated position | Day 15, day 60, day 90, day 120, day 150, day 180
  Assessment of pain related to the semi-seated position using a Visual Analogue Scale (VAS)
Assessment of disorders in falling asleep and sleep quality (micro arousals) | Day 15, day 60, day 90, day 120, day 150, day 180
  Assessment of disorders in falling asleep and sleep quality (micro arousals) by a questionnaire
Assessment of risk of falling using the Yoobreath system™ | Day 15, day 60, day 90, day 120, day 150, day 180
  Number of falls
Assessment of the compliance | Day 0, day 15, day 60, day 90, day 120, day 150, day 180
  Reporting of side effects

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No